CLINICAL TRIAL: NCT00002054
Title: A Double-Blind Study To Evaluate the Long-Term Safety and Effectiveness of 60 mg Versus 120 mg of Aerosol Pentamidine in the Prophylaxis of Pneumocystis Carinii Pneumonia in AIDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisons (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 022C; 87-71 (Part C)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Dose-Response Relationship, Drug; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Pentamidine

INTERVENTIONS:
Drug: Pentamidine isethionate

SUMMARY:
To evaluate the safety, tolerability, and description of time to Pneumocystis carinii pneumonia (PCP) for long-term biweekly administration of 1 of 2 doses of aerosol pentamidine when used as a prophylactic agent in patients who have had one episode of AIDS-associated PCP.

ELIGIBILITY:
Inclusion Criteria

Patients who have completed 16 treatments under Fisons study no. 87-71 entitled, "A Double-Blind Group Comparative Study To Evaluate the Safety and Effectiveness of Three Different Doses of Aerosol Pentamidine in the Prophylaxis of Pneumocystis Carinii Pneumonia in Patients With AIDS Post First Episode PCP." Detailed safety parameters must have been documented for 6 months.

* Patients must receive the first dose on this study within 2 weeks of their last dose under study no. 87-71.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Requiring ongoing active therapy for an opportunistic infection (O.I.) at time of entry or those patients with either of the following AIDS-defining O.I.'s at entry:
* Toxoplasmosis.
* Cryptococcosis.
* Pulmonary Kaposi's sarcoma.
* Asthma poorly controlled by medication.
* Receiving active therapy for tuberculosis.

Patients with the following are excluded:

* Requiring ongoing active therapy for an opportunistic infection (O.I.) at time of entry or those patients with either of the following AIDS-defining O.I.'s at entry:
* Toxoplasmosis.
* Cryptococcosis.
* Pulmonary Kaposi's sarcoma.
* Unwilling to sign informed consent.
* Cannot cooperate with study procedures.
* Asthma poorly controlled by medication.
* Receiving active therapy for tuberculosis.

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Fisons Corp, Rochester, New York, United States

REFERENCES:
- [Background] Hogan CH, Hodges JS, Mugglin A, Peterson PM, Abrams DI, Saravolatz L. The perils of visit-driven endpoints in antiretroviral trials. Int Conf AIDS. 1996 Jul 7-12;11(1):237 (abstract no TuB522)
- [Background] Wulfsohn M, Fischl M, Tsiatis A. Predictors of survival among patients with AIDS receiving zidovudine. Int Conf AIDS. 1992 Jul 19-24;8(2):C314 (abstract no PoC 4419)
- [Background] De Gruttola V, Wulfsohn M, Fischl MA, Tsiatis A. Modeling the relationship between survival and CD4 lymphocytes in patients with AIDS and AIDS-related complex. J Acquir Immune Defic Syndr (1988). 1993 Apr;6(4):359-65. PMID 8095980
- [Background] Lavelle J, Murphy R, Harding P, Pierce P. Aerosolized pentamidine prophylaxis following Pneumocystis carinii pneumonia in patients with AIDS. Int Conf AIDS. 1990 Jun 20-23;6(2):374 (abstract no 2083)